CLINICAL TRIAL: NCT01720498
Title: The Effect Site Concentration of Remifentanil for Preventing QTc Interval Prolongation During Intubation Under Propofol-remifentanil Anesthesia in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Clinical assistant professor, Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0581
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: General Surgery With Endotracheal Intubation
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Male (Experimental): To find out the effect site concentration of remifentanil for preventing QTc prolongation < 15 sec during intubation : Dixon's up-and-down method
  Interventions: Drug: remifentanil
- Female (Experimental): To find out the effect site concentration of remifentanil for preventing QTc prolongation < 15 sec during intubation : Dixon's up-and-down method
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — The effect site concentration of remifentanil

SUMMARY:
To find out the effect site concentration of remifentanil for preventing QTc interval prolongation during intubation under propofol-remifentanil anesthesia in elderly patients

DETAILED DESCRIPTION:
The increase of Corrected QT (QTc) interval is associated with age. It is known that most inhalation anesthetics or intravenous anesthetics can influence the QTc. In addition, tracheal intubation during induction can stimulates sympathetic activity, which, as a results, prolong the QTc interval. Therefore, the aim of study is to find out the effect site concentration of remifentanil for preventing QTc interval prolongation during intubation under propofol-remifentanil anesthesia in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years ASA class I-II who received surgery with endotracheal intubation

Exclusion Criteria:

* emergency surgery
* electrocardiography abnormality
* hypertension
* diabetes mellitus
* end stage renal disease
* moderate to severe cardiac disease
* moderate to severe liver dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The effect site concentration for preventing QTc interval prolongation | 2 min

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea